CLINICAL TRIAL: NCT02419443
Title: The Impact of Perioperative Gabapentin on Chronic Groin Pain After Inguinal Hernia Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew Hannon, CDR, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMCSD.2010.0123
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Peripheral Nerve Disorder Associated With Repair of Hernia
Keywords: inguinal hernia repair, chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients randomized to the placebo-group were administered placebo-pills orally one hour prior to surgery, then three times a day for a maximum of 6 total doses.
  Interventions: Drug: Placebo
- Gabapentin (Active Comparator): Patients randomized to the gabapentin-group were administered 300 mg orally one hour prior to surgery, then three times a day for a maximum of 6 total dose.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Gabapentin is a structural analogue of GABA that decreases activation of voltage-activated calcium channels which may decrease release of excitatory neurotransmitters such as glutamate. Its analgesic mechanisms have been utilized effectively for the treatment of chronic pain in several disorders such as cancer, fibromyalgia and diabetic peripheral neuropathy.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo — Control group
  Arms: Placebo

SUMMARY:
A common source of morbidity after IHR is chronic groin pain(CGP), usually defined as pain lasting longer than 3 months. Gabapentin is an anticonvulsant that is also of benefit in the treatment of neuropathic pain. We propose a randomized, double-blind, placebo controlled study of the effect of gabapentin on CGP after IHR. Their pain will be assessed with a visual analogue scale. For those reporting pain, the need for pain medication, or other treatment, and the effect of pain on their quality of life will be recorded.

DETAILED DESCRIPTION:
Over 500,000 inguinal hernia repairs(IHR) are performed in the United States annually. This is also one of the most common operations performed on the primarily young, male Active Duty population. A common source of morbidity after IHR is chronic groin pain(CGP), usually defined as pain lasting longer than 3 months. The incidence of CGP varies widely in published reports, but in the majority it is 25 to 30%. A major etiology of CGP is thought to be injury to inguinal nerves during surgery. Gabapentin is an anticonvulsant that is also of benefit in the treatment of neuropathic pain. Numerous studies have shown that gabapentin can decrease perioperative pain in patients undergoing surgeries such as hysterectomy, cholecystectomy and spine surgery. Doses and medication regimens varied in these studies, One study in patients undergoing IHR who received a single dose of gabapentin preoperatively, showed a decrease in postoperative pain and in reported pain scores in the first 6 months. We propose a randomized, double-blind, placebo controlled study of the effect of gabapentin on CGP after IHR. Patients will be given placebo or gabapentin. Those given gabapentin, will be given 300 mg orally three times daily for a total of six doses with the first dose given on the morning of surgery. Patients will be evaluated preoperatively and at 1, 6, 12 and 24 months after surgery. Their pain will be assessed with a visual analogue scale. For those reporting pain, the need for pain medication, or other treatment, and the effect of pain on their quality of life will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18 years of age or older undergoing initial inguinal (bilateral or unilateral) hernia repair by any method (i.e. laparoscopic or open surgery)

Exclusion Criteria:

* Age less than 18 years of age, recurrent hernias, emergency operations, already taking gabapentin, allergy to gabapentin, pre-existing chronic pain or psychiatric disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Pain score | 24 months
  Visual analog scale

SECONDARY OUTCOMES:
Quality-of-life (QOL) | 24 months
  SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hannon, M.D., Principal Investigator — United States Naval Medical Center, San Diego

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated results will be made available.

REFERENCES:
- [Background] Poobalan AS, Bruce J, Smith WC, King PM, Krukowski ZH, Chambers WA. A review of chronic pain after inguinal herniorrhaphy. Clin J Pain. 2003 Jan-Feb;19(1):48-54. doi: 10.1097/00002508-200301000-00006. PMID 12514456
- [Background] van Hanswijck de Jonge P, Lloyd A, Horsfall L, Tan R, O'Dwyer PJ. The measurement of chronic pain and health-related quality of life following inguinal hernia repair: a review of the literature. Hernia. 2008 Dec;12(6):561-9. doi: 10.1007/s10029-008-0412-y. Epub 2008 Aug 21. PMID 18716856
- [Background] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Background] Kong VK, Irwin MG. Gabapentin: a multimodal perioperative drug? Br J Anaesth. 2007 Dec;99(6):775-86. doi: 10.1093/bja/aem316. PMID 18006529
- [Derived] Quail J, Spence D, Hannon M. Perioperative Gabapentin Improves Patient-Centered Outcomes After Inguinal Hernia Repair. Mil Med. 2017 Nov;182(11):e2052-e2055. doi: 10.7205/MILMED-D-17-00107. PMID 29087880